CLINICAL TRIAL: NCT04353050
Title: A Multicenter, Ambispective, Low-interventional Clinical Study Evaluating Molecular Genetic Markers for Non-invasive Differential Diagnosis of Benign and Malignant Pigmented Skin and Mucosal Neoplasms
Brief Title: Atypical MOLes and Melanoma Early Detection Study (MoleMed)
Acronym: MoleMed
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Russian Academy of Medical Sciences (Other)
Collaborators: Blokhin's Russian Cancer Research Center (Other)
Responsible Party: Principal Investigator, Igor Samoylenko, Principal Investigator, Senior Researcher, Department of Oncodermatology, MD, PhD, Blokhin's Russian Cancer Research Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MoleMed-0320
Record Dates: First submitted 2020-04-13; First posted 2020-04-20 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Melanoma; Melanoma (Skin); Moles; Nevus; Nevus, Blue; Nevus, Pigmented; Nevus, Spitz; Nevi, Spindle Cell; Nevi, Dysplastic; Dysplastic Nevus Syndrome; Mucosal Melanoma; Mucosal Melanosis
Keywords: non-invasive diagnosis; melanoma; atypical moles; dysplastic nevi
MeSH Terms: conditions — Melanoma; Nevus; Nevus, Blue; Nevus, Pigmented; Nevus, Epithelioid and Spindle Cell; Nevus, Spindle Cell; Dysplastic Nevus Syndrome | interventions — Transdermal Patch

STUDY DESIGN:
Intervention Model Description: Ambispective study with two retrospective cohorts and one prospective cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (retrospective) (No Intervention): Only data from medical records and formalin-fixed paraffin-embedded tissue blocks will be collected from patients in this cohort. Patients with skin or mucosal melanoma and dysplastic nevi which have been already excised are eligible. FFPE tissue blocks with MPATH-Dx Class 1-2 vs Class 3-5 will be collected in approximately 1:1 ratio
- Cohort 2 (retrospective) (No Intervention): Only data from medical records, formalin-fixed paraffin-embedded tissue blocks and cytologic slides will be collected from patients in this cohort. Patients with skin or mucosal melanoma and dysplastic nevi which have been already excised are eligible. FFPE tissue blocks with MPATH-Dx Class 1-2 vs Class 3-5 will be collected in approximately 1:1 ratio
- Cohort 3 (prospective) (Other): Patients with pigmented lesions on the skin or mucosa who are referred for excisional biopsy will be offered to apply investigated non-invasive adhesive system on their lesion just before the excisional biopsy. After biopsy cytological slides and FFPE tissue blocks will be prepared. All three types of obtained samples will be investigated separately (adhesive patches, cytologic slides and FFPE tissue blocks) for genetic markers whereas cytologic slides and FFPE tissue blocks will be processed also routinely and regular cytologic and histopathologic report will be generated.
  Interventions: Procedure: Non-invasive adhesive system (patch)

INTERVENTIONS:
Procedure: Non-invasive adhesive system (patch) — The already registered on the market adhesive skin patch will be applied and removed for several times on the pigmented skin (or mucosal) lesion just before the preplanned excisional biopsy after local anaesthesia have been already administered. Excisional biopsy and local anaesthesia are not the part of this study and will be carried out according to local practice
  Arms: Cohort 3 (prospective)

SUMMARY:
This is a multicenter, ambispective, low-interventional clinical study evaluating molecular genetic markers for non-invasive differential diagnosis of benign and malignant pigmented skin and mucosal neoplasms. In retrospective cohorts genetics markers will be identified. In prospective cohort non-invasive adhesive system will be tested to identify malignant or benign lesions with prespecified sensitivity and specificity compared to other non-invasive techniques (i.e. dermoscopy) and using histopathological examination as a "golden standard".

ELIGIBILITY:
Inclusion Criteria:

Cohort 1 (retrospective):

* Histologically confirmed diagnosis of melanocytic neoplasm of the skin or mucous membranes (benign, malignant or with unclear potential);
* The presence of a paraffin block with a tumor suitable for molecular genetic analysis;
* Signed informed consent form for living patients (for deceased, signing of a consent form with legal representatives is not required);
* Patient's age is over 18 years for the period of inclusion in the study (at the time of signing the consent form for living patients or for the excision biopsy period for deceased patients);
* Known clinical data of the patient (gender, age, skin phototype), hereditary history, medical history and follow-up of treatment outcomes for at least 5 years

  2. Cohort 2 (retrospective):
* Histologically confirmed diagnosis of melanocytic neoplasm of the skin or mucous membranes (benign, malignant or with unclear potential);
* The presence of a paraffin block with a tumor suitable for molecular genetic analysis
* The presence of cytological preparations (at least 2 glasses) of the primary tumor with tumor material
* Signed informed consent form for living patients (for deceased, signing of a consent form with legal representatives is not required);
* Patient's age is over 18 years for the period of inclusion in the study (at the time of signing the consent form for living patients or for the excision biopsy period for deceased patients);
* A known medical history and follow-up of treatment outcomes for at least 6 months.

  3. Cohort 3 (prospective):
* Clinically (including any type of dermatoscopy or other non-invasive diagnostic methods) suspected diagnosis of malignant melanocytic neoplasm (or neoplasms) of the skin or mucous membranes (or lesion(s) with unclear malignant potential)
* The patient is scheduled to undergo an excision biopsy (or wide excision) of the neoplasm (s) of the skin or mucous membranes within 3 months from the date of inclusion in the study and the patient is able to tolerate this intervention;
* Signed Informed Consent Form

Exclusion Criteria:

Cohort 1:

* Unknown histological diagnosis (no information on the melanocytic nature of the neoplasm)
* Unsuitable for analysis paraffin block with a tumor or its absence
* Unknown history or lack of traceability after diagnosis within 5 years
* For the period of inclusion in the study (signing an informed consent form for living patients or an excision biopsy for deceased patients), the patient's age is under 18 years

  2. Cohort 2:
* Unknown histological diagnosis (no information on the melanocytic nature of the neoplasm)
* Unsuitable for analysis paraffin block with a tumor or its absence
* Unsuitable for analysis cytological preparations/smears (or the absence of tumor cells in cytological preparations)
* Unknown history or lack of traceability after diagnosis within 6 months.
* For the period of inclusion in the study (signing an informed consent form for living patients or an excision biopsy for deceased patients), the patient's age is under 18 years

  3. Cohort 3 (prospective):
* The patient is NOT scheduled to undergo an excision biopsy (or wide excision) of the neoplasm (s) of the skin or mucous membranes in the next 3 months since inclusion in the study OR the patient is not able to tolerate this intervention;
* The available morphological or cytological confirmation of the nature of the neoplasm (s) (benign or malignant), which (s) is planned to be removed in the framework of this study,
* Ulcerated neoplasms;
* Contact bleeding neoplasms;
* Non-melanocytic neoplasms;
* Neoplasms with an area of more than 5 sq. cm
* Neoplasms located subcutaneously or in soft tissues and, according to clinical signs, not associated with the skin
* Known allergy to any component of the applied adhesive system;
* Inability of the patient to follow the study procedures (including contacting the researcher during the follow-up visits) or other reasons that, in the opinion of the principal investigator, may become an obstacle for the patient to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity on the investigated non-invasive genetic method for diffrential diagnosis of benign and malignant melanocytic lesions compared to histopathological examination | April 2020 - Nov 2022
  •Assessment of the sensitivity and specificity of a complex of molecular genetic studies applicable for non-invasive differential diagnosis of benign and malignant melanocytic neoplasms of the skin and mucous membranes in comparison with a standard histological examination

SECONDARY OUTCOMES:
Sensitivity and specificity on the investigated non-invasive genetic method for diffrential diagnosis of benign and malignant melanocytic lesions compared to other non-invasive diagnostic tools (i.e. dermoscopy) | up to 12 months
  Assessment of the sensitivity, specificity, positive and negative prognostic significance of the developed molecular genetic method for non-invasive differential diagnosis of benign and malignant pigmented neoplasms of the skin and mucous membranes in comparison with clinical diagnosis with an naked eye by an oncologist or dermatologist
Describe some parameters of the identified malignant tumors | up to 12 months
Describe the frequency of relapse (local, regional and systemic) within the observation period | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Igor V Samoylenko, MD, PhD, Principal Investigator — N.N. Blokhin Russian Cancer Research Center of Russian MoH
Locations (2):
- Russia (2):
  - N.N. Blokhin Russian Cancer Research Center, Moscow, Moscow
  - Privolzhsky Research Medical University of the Ministry of Health of the Russian Federation, Nizhny Novgorod

IPD SHARING:
Plan to Share IPD: No